CLINICAL TRIAL: NCT04362904
Title: Acupressure for Cancer Related Fatigue in Elderly Cancer Patients: A Randomized Controlled Study
Brief Title: Acupressure for Fatigue in Elderly Cancer Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: TC Erciyes University (Other)
Responsible Party: Principal Investigator, ülkü özdemir, assistant professor doctor, TC Erciyes University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: TDK-2014-5025
Record Dates: First submitted 2020-04-17; First posted 2020-04-27 (Actual); Last update posted 2020-04-27 (Actual); Status verified 2020-04

CONDITIONS: Fatigue
Keywords: Acupressure; Cancer; Fatigue; Elderly individuals; Nursing
MeSH Terms: conditions — Fatigue; Neoplasms | interventions — Acupressure

STUDY DESIGN:
Intervention Model Description: a randomized, controlled trial in pre-test post-test design
Oversight: Data Monitoring Committee: No

ARMS (2):
- acupressure (Experimental): In accordance with the acupressure protocol, each day for four weeks, taking into account the awakening and sleep periods of the individuals, acupressure applied for a total of 3 min to the each acupuncture points (one session 18 minutes) twice a day between 07:00 and 10:00 and 19:00 to 22:00 in the morning patients were asked to perform acupressure by their caregivers or on their own.
  Interventions: Other: acupressure
- control (No Intervention): No intervention was applied to the control group.

INTERVENTIONS:
Other: acupressure
  Arms: acupressure

SUMMARY:
The aim of this study was to investigate the effect of acupressure on the severity and level of cancer-related fatigue in elderly patients with cancer.

DETAILED DESCRIPTION:
Participants The research was carried out in two stages: quantitative and qualitative. The quantitative phase of the study was a randomized, controlled trial in pre-test post-test design. The second phase of the study was performed as a qualitative study by using individual in-depth interview method at the end of four weeks of acupressure.

The study was conducted with the volunteers from hematology and medical oncology clinic in a university hospital, in Turkey.

At the beginning of the study, a total of 20 patients, 10 for each acupressure and control groups, were included in order to calculate the sampling size of the study. As the result of the evaluation, a total of 28 patients (14 for acupressure, 14 for control groups) with 95% confidence level and 90% strength were included in the study. It was decided that 11 patients would be added to both group to reach the total of 50 patients (25 acupressure group, 25 control group) considering withdrawals from the study. Acupressure and control groups were randomized by computerized patient selection. The study was completed with a total of 31 patients (15 acupressure, 16 control group) who met the inclusion criteria At the end of the study, 95% confidence level was found as 99% for Visual Analog Scale (VAS) and 95% for total Piper Fatigue Scale (PFS) score in acupressure and control groups.

In order to carry out the study, the permission of the Ethics Committee of the Clinical Researches (decision no: 2013/670) and written permission was received from the clinics where the study will be conducted. The study was carried out in accordance with the provisions of the Declaration of Helsinki (1995). Written informed consent was obtained from each participant.

In the qualitative phase of the study, in-depth interviews with individuals in the acupressure group were recorded with a voice recorder.

Procedure Routine treatment of the patients, added in the acupressure and control groups according to inclusion criteria, was not intervened during the study.

In order to collect the pre-test data of the patients in the acupressure group and the control group in the begining, the PFS researcher administered the patient identification form, VAS, by face-to-face interviews with the patients.

For this study, studies on literature are examined and acupressure application protocol was prepared by getting an expert opinion.

The researcher who applied acupressure participated in an acupressure course for 8 hours of training of acupuncture points and acupressure application including 4 hours of acupressure technique training.

In acupressure application, each acupuncture point was applied with acupressure device (Acu-Doctor Electro Acupuncture Device LY508). The device includes a digital display for acupuncture point location and a button for stimulating the acupuncture point after spot detection.

At the end of four weeks, VAS and PFS applied to the all patients again. In the qualitative phase of the study, the researcher took experience and opinions of the patients in the acupressure group about acupressure application during the second follow-up period. In the in-depth interview, a semi-structured Acupressure Experience Patient Opinion Form includes questions about acupressure was applied.

Preliminary Application In order to determine the operability of the Patient Introduction Form, acupressure application and its duration and the applicability of the scales 5 elderly patients with cancer were pre-treated with the acupressure. Pre-application data were excluded from the research.

Intervention Acupressure Group: For acupressure application, three acupuncture points (Liver 4 (LI4), Stomach 36 (ST36), Spleen 6 (SP6)) on both hands and legs are selected by taking expert advice and based on previous fatigue studies. The point LI4 corresponds to the midpoint between the first and second carpal bones. It is in the middle of the second metacarpal bone on the radial side. The ST36 point is located below the tibia, approximately 4 finger wide, along the outer edge of the tibia and 1.5-2 finger apart from the tibia, above the anterior tibia muscle. SP6 is located on the spleen meridian, on the inner side of the lower leg, 4 fingers above the ankle, behind the tibia. It is on the caudal edge of the tibia, three units in the proximal of the medial malleolus end region.

The acupuncture points, acupressure to be applied, were determined by the researcher at the first interview, by measuring the patients' own finger measurements and also by the acupressure device. The zones are then marked with an indelible pen. Then, the researcher in accordance with the acupressure protocol trained all the patients in the acupressure group or the individuals responsible for the care of the patients. After the participants were observed while performing acupressure correctly and after making them comfortable in all steps, the patients were given an application-training guide prepared by the researcher. The contents of the guide include information on acupuncture points and acupressure application. The participants were given a stopwatch to adjust the time with the acupressure device. In accordance with the acupressure protocol, each day for four weeks, taking into account the awakening and sleep periods of the individuals, acupressure applied for a total of 3 min to the each acupuncture points (one session 18 minutes) twice a day between 07:00 and 10:00 and 19:00 to 22:00 in the morning patients were asked to perform acupressure by their caregivers or on their own. All participants were monitored weekly by telephone.

The determined intensity, frequency and sensitivity were noted for each patients and recorded on the Patient Monitoring Chart - Patient Form. It is explained that for each acupuncture point, the procedure will start from head towards feet and the right hand side, then will continue with the point on the left side before moving to a different point. The patients were asked to record the acupressure application on the Patient Monitoring Chart-Patient Form. At the first interview, the Patient Presentation Form and the other scales were applied which took approximately 20 minutes, and the acupressure training lasted an average of 45 minutes.

The in-depth interviews conducted by the researcher at the end of the acupressure application were conducted in a suitable room in the hospital or in the patients' own homes. During the interviews, the patients' experiences were recorded with a voice recorder after obtaining the permission of the patients. Interviews took an average of 10 to 15 minutes.

Control Group: No intervention was applied to the control group.

ELIGIBILITY:
Inclusion Criteria:

* Age 65 and over
* Who completed chemotherapy treatment for cancer at least a month ago
* Least literate
* Moderate to severe fatigue (VAS fatigue score 4 and above)
* Platelet count> 50,000
* Hemoglobin levels> 9 g / dl
* Hematocrit levels> 30%
* Patients with an estimated survival time of more than three months

Exclusion Criteria:

* Comorbidities that may cause fatigue (eg moderate and severe heart failure, hypothyroidism, diabetes, multiple sclerosis)
* Being diagnosed with a psychiatric disease
* Nerve, soft tissue and vascular disease on acupressure areas (hand and leg)
* Infection and surgery operations on acupressure areas (hand and leg)
* Patients had chemotherapy, radiotherapy or other cancer treatment planned during the study

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 31 (Actual)
Dates: Start 2014-08-04 (Actual); Primary Completion 2016-03-10 (Actual); Study Completion 2016-03-10 (Actual)

PRIMARY OUTCOMES:
Visual Analog Scale | four weeks
  The scale is a 10-cm scale starts with a -0- representing "I don't feel tired", the other end is -10- "I feel very tired". 0-3 points show mild fatigue, 4-6 points moderate fatigue, 7-10 points indicate severe fatigue. The patients were asked to mark how tired they were during the last week on a scale of 0 to 10. The distance between the marked point and the lowest end of the line (0 = no fatigue) was measured in centimeters by the ruler and the numerical value was determined as the fatigue score of the patients.
Piper Fatigue Scale | four weeks
  The scale evaluates the patient's subjective perception of fatigue with four sub-dimensions. These sub-dimensions are behavioral/severity sub-dimension that evaluates effects and intensity of fatigue on daily life activity (DLA), affective meaning sub-dimension that includes emotional meaning attributed to fatigue, sensory sub-dimension that reflects spiritual, physical and emotional symptoms of fatigue and cognitive/mood sub-dimension that reflects the level of effects of fatigue on cognitive functions and state of mind. The high scores obtained from the scale indicate that the perceived fatigue level is high.The validity and reliability study of the scale for the Turkish population was conducted by Can and the cronbach alpha coefficient was found to be 0.94. The cronbach's alpha coefficient in this study was 0.79 in the first follow-up and 0.94 in the second follow-up.

OTHER OUTCOMES:
Acupressure Experience Patient Opinion Form | four weeks
  In the qualitative phase of the study, the was used during in-depth interviews with the individuals in the acupressure group at the end of four weeks of acupressure application. It was developed as semi-structured interview by the researcher to learn the experiences and opinions of individuals. The form includes questions about acupressure (effects of acupressure, effects of fatigue, easy and difficult aspects of the application, whether to recommend acupressure application for fatigue).

CONTACTS AND LOCATIONS:
Overall Officials: ülkü özdemir, Principal Investigator — TC Erciyes University; sultan taşcı, Study Director — TC Erciyes University

IPD SHARING:
Plan to Share IPD: No
no panning